CLINICAL TRIAL: NCT06682104
Title: Individual Intensive Short Term Psychodynamic Psychotherapy for Patients with Treatment Resistance Persistent Physical Symptoms
Brief Title: ISTDP for Patients with Treatment Resistance PPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Maroti (Other)
Responsible Party: Sponsor-Investigator, Daniel Maroti, PhD, principal investigator, Stockholm University
Organization: Stockholm University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOSMOS3-Individual ISTPD
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Somatic Symptom Disorder; Persistent Physical Symptoms; Functional Somatic Syndrome; Functional Somatic Disorder; Medically Unexplained Symptoms
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individual intensive short term psychodynamic therapy (Other): The Individual Intensive Short-Term Psychodynamic Psychotherapy (ISTDP) arm for patients with Persistent Physical Symptoms (PPS) focuses on addressing the underlying emotional and psychological factors contributing to these chronic symptoms. In this treatment arm, participants engage in structured, one-on-one psychotherapy sessions with a trained ISTDP therapist.
  Interventions: Behavioral: Individual intensive short term psychodynamic therapy

INTERVENTIONS:
Behavioral: Individual intensive short term psychodynamic therapy — ISTDP aims to help patients explore and process unconscious emotions, particularly those linked to past trauma or unresolved conflicts, that may be contributing to their physical symptoms. Patients are guided to identify and express repressed feelings such as anger, grief, or fear. The therapist actively engages the patient in a focused and intensive manner, helping them to recognize emotional defenses, break through resistance, and experience these emotions directly in the therapeutic setting.

SUMMARY:
Intensive Short-Term Psychodynamic Psychotherapy (ISTDP) for Treatment-Resistant Persistent Physical Symptoms is a therapeutic approach designed to help patients whose physical symptoms have not responded to traditional medical or psychological treatments. These persistent physical symptoms (PPS) often include conditions such as chronic pain, fatigue, or gastrointestinal issues, where a psychological component may be involved.

ISTDP focuses on identifying and addressing unconscious emotional conflicts, which are thought to contribute to or exacerbate physical symptoms. The therapy encourages patients to recognize and express repressed emotions, such as anger, sadness, or fear, which may manifest somatically if left unresolved.

For patients with treatment-resistant PPS, ISTDP offers a focused, time-limited intervention aimed at breaking the cycle of emotional suppression and physical symptomatology. The method involves intense therapeutic engagement, fostering a direct experience of emotions in a controlled environment. Through this process, patients often gain emotional awareness and experience symptom relief.

Research on ISTDP in this population suggests that it can effectively reduce the severity of physical symptoms, improve emotional well-being, and enhance overall functioning when other treatments have not yielded significant results.

For patients with treatment-resistant PPS, ISTDP offers a focused, time-limited intervention aimed at breaking the cycle of emotional suppression and physical symptomatology. The method involves intense therapeutic engagement, fostering a direct experience of emotions in a controlled environment. Through this process, patients often gain emotional awareness and experience symptom relief.

Research on ISTDP for this population suggests that it can be effective in reducing the severity of physical symptoms, improving emotional well-being, and increasing overall functioning when other treatments have failed to produce significant results.

ELIGIBILITY:
Inclusion Criteria:

* The participant certifies that they have undergone a medical evaluation for their physical symptoms.
* The participant rates either moderate distress from physical symptoms on the PHQ-15 form (over 10 points) or significant distress from a single physical symptom (at least 2 points for that symptom).
* The participant expresses interest in exploring whether emotional factors, such as stress, may contribute to their symptom profile.
* Any prescribed medications must have been stable for at least 1 month.
* Participants must meet the criteria for non-response/treatment resistance, i.e., no reliable change in PHQ-15.

Exclusion Criteria:

* Participants suffer from ongoing substance abuse (alcohol or drugs) or are assessed to have severe mental health issues (psychotic disorders, moderate to high suicide risk, antisocial personality disorder, etc.).
* Participants are currently prescribed medications that are clearly addictive and sedative in nature (e.g., benzodiazepines).
* Participants are involved in other psychological treatments focused on physical symptoms. However, other psychological treatments are allowed as long as the supportive therapy does not occur more than once a month.
* Participants do not have sufficient proficiency in the Swedish language.
* Somatic symptoms is judged to be need further medically evaluation or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionaire-15 (PHQ-15) | Lineal regression model using measurement points from from pre-treatment, 1 week before treatment and during treatment (up to 5 months)
  Somatic symptom severity during the "last week" was assessed with the PHQ-15. Items were rated 0 ("Not bothered at all"), 1 ("Bothered a little"), or 2 ("Bothered a lot"); total scores range from 0 to 30 for women and 0-27 for men.
Visual Analoge Scales | Lineal regression model using measurement points from from pre-treatment, 1 week before treatment and during treatment (up to 5 months)
  Visual Analoge Scales suggested by the EURONET-SOMA network (Rief et al., 2017). Somatic symptom intensity was measured from 1 ("No symptom") to 10 ("Symptom as bad as you can imagine") and somatic symptom interference from 1 ("No interference") to 10 ("Maximum interference").

SECONDARY OUTCOMES:
Patient Health Questionaire-9 (PHQ-9) | Measured before treatment start and post treatment (after 16 weeks of treatment).
  PHQ-9 consists of nine questions withs ratings 0-3 (0= "not at all", 3= "almost every day") on impact of depressive symptoms. Higher scores indicate worse symptom/functioning with a maximum score of 27.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Measured before treatment start and post treatment (after 16 weeks of treatment).
  GAD-7 consists of seven questions with ratings 0-3 (0= "not at all", 3= "almost every day") on impact of anxiety symptoms. Higher scores indicate worse symptom/functioning functioning with a maximum score of 21.
Post traumatic symptom Check List-5 (PCL-5) | Measured before treatment start and post treatment (after 16 weeks of treatment).
  PCL-5 consists of 20 questions with ratings 0-4 on impact of post traumatic symptoms. Higher scores indicate worse symptom/functioning with a maximum score of 80.

OTHER OUTCOMES:
Negative Effects Questionnaire (NEQ) | At post-treatment (after 16 weeks of treatment)]
  Participants respond to a series of statements regarding potential negative effects they may have experienced during or after therapy, typically using a Likert scale (e.g., 1 = "Not at all," to 5 = "Extremely"). The total score is computed by summing the responses, where higher scores indicate a greater frequency or severity of negative effects.
Patient Session rating scale (with 8 additional questions) | Each week once a week throughout 16 weeks of treatment
  Session Rating Scale (SRS) evaluates the therapeutic alliance and the quality of the therapy session. It consists of four items rated on a scale from 0 ("Not at all") to 10 ("Extremely") that assess various aspects of the therapy session, including the therapist's understanding of the patient, the relevance of the session, the connection between the patient and therapist, and how well the patient's needs were addressed. In the same manner 8 additional questions on experienced emotions are asked (e.g. on a scale 0-10 how much shame was experienced in the therapy session).
Therapist Rating after each ISTDP session | Each week once a week throughout 16 weeks of treatment
  "Therapist Rating after each ISTDP session" measures several aspects of the therapeutic process and the patient's emotional response during the session. For example, on a five point Likert scale - To a very small extent" to "To a very high extent - the therapist rate the extent to which he/she focused on and/or used typical ISTDP interventions during the session.
Patient Health Questionaire-4 (PHQ-4) | Each week once a week throughout 16 weeks of treatment
  PHQ-4 consists of four questions withs ratings 0-3 (0= "not at all", 3= "almost every day") on impact of depressive symptoms. Higher scores indicate worse symptom/functioning with a maximum score of 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm University, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Participants have not approved this.